CLINICAL TRIAL: NCT06740305
Title: NASA Prebreathe Study
Acronym: NASA Prebreath
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Initial funding ended; expect future funding. Will resume recruiting at that time.
Sponsor: Duke University (Other)
Collaborators: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00116846; 80NSSC24PB887 (Other Grant/Funding Number: NASA)
Record Dates: First submitted 2024-11-19; First posted 2024-12-18 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Decompression Sickness
Keywords: Space; Microgravity; Decompression; Decompression sickness; Altitude
MeSH Terms: conditions — Decompression Sickness | interventions — Altitude; Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Healthy Volunteers (Experimental): Each participant in this group will be exposed to simulated altitude.
  Interventions: Other: Altitude; Drug: 100% Oxygen

INTERVENTIONS:
Other: Altitude — Subjects will be exposed to simulated altitude (30,000 ft, 4.3 psia) in a hypobaric chamber. This is the same ambient pressure to which astronauts are exposed during EVA ("space walks").
Drug: 100% Oxygen — Oxygen pre-breathing prior to altitude or simulated high altitude exposure is routinely used by the Air Force, NASA and organizations such as Duke Medical Center to prevent and treat decompression sickness as well as for treatment of patients. Oxygen used for this study is medical grade.

SUMMARY:
This study will validate the experimental method and chamber facility at the Duke Center for Hyperbaric Medicine & Environmental Physiology and test team capabilities to support NASA decompression sickness (DCS) studies. This project is related to development of protocols for extravehicular activity (EVA, "spacewalks") to minimize the risk of decompression sickness. Duke will perform four test days, collecting and recording data each day. Each test day will involve 3 volunteer subjects ages 18-50 years, who will breathe 100% oxygen for 6 hours. This will be followed by 6 hours in the hypobaric chamber at 1/3 atmosphere, during which subjects will perform various tasks, including arm and leg exercises, and undergo ultrasound testing to detect vascular bubbles. End-points will include bubble scores, and decompression sickness (DCS). If subjects develop DCS symptoms they will immediately be recompressed to ambient pressure and be assessed and treated.

DETAILED DESCRIPTION:
Applicants will be screened to provide at least 3 subjects plus one test operator (Doppler /ultrasound technician) per day to participate in four 12-hour chamber runs for this pilot testing. Screening back-up subjects in case of subject availability issues, withdrawal, or disqualification will be included. Subjects will be screened per standard protocols, and the subject pool will include females to demonstrate their capabilities to recruit and test this important population. NASA will provide inclusion and exclusion criteria for a population demographic similar to the astronaut corps. Following a screening process, subjects will participate in a familiarization session during which they will receive verbal and written description of the test protocol, be encouraged to ask questions, and will provide written informed consent before proceeding to participation. Thereafter, subjects will be familiarized with the chamber protocol and safety procedures. Subjects also will be familiarized with the EVA simulation workstations, and metabolic rate will be measured while performing the arm ergometry and stepping exercises at several low work rates (submaximal exercise intensity) to verify the cadence or work rates required for the in-chamber exercise prescription.

A test plan will be implemented that includes a 6-hour prebreathe of 100% oxygen using a transparent hyperbaric hood, followed by a simulation of EVA lasting 6 hours, or until signs and symptoms that require test termination (per NASA and Duke standards), test termination by subject request, or facility or monitoring capabilities malfunctions. These sessions will include successful mask operations and demonstration of safety procedures. An additional 30 minutes will be allotted for re-pressurization and post-test monitoring.

Appropriate medical support will be provided to perform pre-chamber physical examination before ingress, during the protocol, for treatment and management of subjects as needed, clearance of subjects after the protocol is completed, and follow-up in the days after the chamber run, as required. Responsibilities of the medical personnel include monitoring and interpretation of 2-D ultrasound and Doppler as well as monitoring of the subject's self-report and symptoms of DCS or intolerance. Prebreathe Conditions The Duke Center for Hyperbaric Medicine & Environmental Physiology will demonstrate the capability to perform 100% O2 prebreathe durations up to 6 hours. Subjects will begin O2 breathing at the start of the prebreathe and continue breathing 100% O2 through decompression and until re-pressurization is completed. Subjects will be provided fluids ad libitum without a break in prebreathe (using drink port). NASA will provide the breathing masks and/or design for their construction or provide approval for a suitable substitution. Food will be allowed prior to start of mask prebreathe but not during the test protocol (for 12 hours). Subjects also are not allowed to sleep during the test protocol. EVA Simulation Duke will demonstrate their capacity to perform a simulated 6-hour EVA and maintain standardized monitoring practices. To simulate the suit environment, the chamber will depress to 4.3 psia (0.3 ATA, approximately 30,000 ft altitude) before initiating the EVA simulation tasks described below. The start time of the EVA is defined by the arrival at the desired level of decompression, and the end time of the EVA is defined by the start of re-pressurization. EVA simulation will include rotation of each subject through a repetitive series of tasks at predetermined intervals in a pre-determined order using a NASA-defined or provided workstations. The EVA is simulated using eight stations, nominally performed in 2 cycles of 4 stations, with subjects rotating between stations every 5 minutes. In one cycle, subjects will rotate through stations that simulate ambulation (low step), upper body technical tasks (standing board), and load carrying (weight transfer), and 2-D ultrasound while subjects are supine on a cot. In the other cycle, subjects will rotate through stations that simulate more vigorous ambulation (high step), upper body physical exertion (arm ergometry), technical tasks performed in a kneeling position (kneeling board), and Doppler ultrasound while supine. Thus, in each cycle subjects will perform 15 minutes of low- to moderate-intensity exercise followed by 5 minutes of monitoring and rest. Work rates during arm ergometry (cadence and resistance) and stepping (cadence) will be prescribed based upon the results of the VO2pk test and the pre-test EVA simulation familiarization with metabolic gas analysis. During ultrasound imaging and Doppler waveform acquisition, at least 10 cardiac cycles will be monitored and recorded in each of three conditions in sequential order: rest, flexing/bending of the arms and legs, and rest. Compliance of the subjects with the prescribed procedures should be documented, including the time at each station, work rates (cadence and load), symptoms reported by the subjects, and test operator observations.

A standardized set of measurements will be used to monitor and document test subjects during the prebreathe, decompression, and recompression. Test operators will record all symptoms reported by the test subjects throughout the duration of the protocol, whether in response to prompting by the test operators or spontaneous self-reporting. Subjects will be removed from the chamber and repressurized (airlock or chamber) at the onset of DCS (Type I or Type II). NASA defines DCS severity with the following criteria: Mild DCS (Type I), Uncomplicated: Symptoms involving joint pain, peripheral nervous system, or simple skin bends that resolve upon repress or within the first 20 minutes of treatment. Mild DCS (Type I), Complicated: Symptoms involving joint pain, peripheral nervous system, or simple skin bends that DO NOT resolve upon repress or within the first 20 minutes of treatment. Mild DCS (Type I) - Repetitive: Mild DCS symptoms involving joint pain, peripheral nervous system, or simple skin bends that occur after a successful treatment and within 30 days of a prior case of DCS for ground-based exposure. These are considered discrete occurrences of DCS in response to chronologically discrete exposures. Serious DCS (Type II): Symptoms involving the Central Nervous System (CNS), cardiovascular system (circulatory collapse/shock), pulmonary system (chokes).

Test operators will query subjects for responses to standardized questionnaires during each rotation through the resting/ultrasound station. Subjects will report a rating of perceived exertion (RPE) and pain using NASA-defined scales at the end of each exercise bout (i.e., after 5 minutes of arm ergometry, stepping).

2-D imaging and Doppler ultrasound for detection of venous gas emboli will be performed by a qualified test operator during each rotation through the resting/ultrasound station while the subject is at rest and following exercise. Doppler and 2-D ultrasound will be recorded and stored electronically with relevant metadata (e.g., subject ID) for post-exposure review and analysis. Doppler results will be scored using the Spencer coding convention and ultrasound will be scored using the Eftedal-Brubbak (EB) scale (0-7).

Heart rate will be continuously monitored and recorded from which data can be downloaded and stored electronically for post-exposure analysis. Test operators will be able to observe the current heart rate from the device as needed and will manually record heart rate at the end of each 5-minute rotation through the EVA simulation stations.

Oxygen saturation (SpO2) will be monitored and recorded continuously during the prebreathe, decompression, and recompression using a device from which the data can be downloaded and stored electronically for post-exposure analysis. Test operators must be able to observe the current SpO2 from the device as needed and will manually record SpO2 at the end of each 5-minute rotation through the EVA simulation stations.

At the conclusion of each test day, Duke will deliver electronic records to NASA using a secure, NASA approved method. The data package will include subject metadata, console and/or operator's logs (including chamber event time, prebreathe records, EVA time, EVA station schedule), chamber pressure recordings (demonstrating depress and repress rates as well as sustained chamber pressure), chamber environmental conditions (partial pressures of O2, CO2, and N2, temperature, humidity), questionnaires, medical monitoring logs, heart rate and pulse oximetry records (if recorded), Doppler and ultrasound recordings, in-chamber video of EVA workstations, and DCS case descriptions. Doppler and ultrasound images will be scored by 3 reviewers in a blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers
* VO2pk >35 ml/kg/min (males)
* VO2pk >30 ml/kg/min (females)

Exclusion Criteria:

* Pregnancy
* Lung and heart disease
* Hypertension
* Diabetes
* Musculoskeletal pain conditions
* Need for regular medications such as analgesics

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with each type of decompression sickness | 24 hours
  Mild DCS (Type I), Uncomplicated: Symptoms involving joint pain, peripheral nervous system, or simple skin bends that resolve upon repress or within the first 20 minutes of treatment.
  Mild DCS (Type I), Complicated: Symptoms involving joint pain, peripheral nervous system, or simple skin bends that DO NOT resolve upon repress or within the first 20 minutes of treatment.
  Mild DCS (Type I) - Repetitive: Mild DCS symptoms involving joint pain, peripheral nervous system, or simple skin bends that occur after a successful treatment and within 30 days of a prior case of DCS for ground-based exposure. These are considered discrete occurrences of DCS in response to chronologically discrete exposures.
  Serious DCS (Type II): Symptoms involving the Central Nervous System (CNS), cardiovascular system (circulatory collapse/shock), pulmonary system (chokes).

SECONDARY OUTCOMES:
Number of participants with venous gas embolism | 24 hours
  Ultrasound will be used to detect circulating bubbles

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Moon, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mollerlokken A, Blogg SL, Doolette DJ, Nishi RY, Pollock NW. Consensus guidelines for the use of ultrasound for diving research. Diving Hyperb Med. 2016 Mar;46(1):26-32. PMID 27044459
- [Background] Le DQ, Dayton PA, Tillmans F, Freiberger JJ, Moon RE, Denoble P, Papadopoulou V. Ultrasound in decompression research: fundamentals, considerations, and future technologies. Undersea Hyperb Med. 2021 First Quarter;48(1):59-72. doi: 10.22462/01.03.2021.8. PMID 33648035
- See also: Related Info — https://sam.gov/opp/e342e7c8ccbe453890a56176d6f2b48d/view

DOCUMENTS (1):
  • Informed Consent Form (2025-06-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT06740305/ICF_000.pdf